CLINICAL TRIAL: NCT06399250
Title: Three Channel Food Concept: the Effect on Food Intake During Hospitalization (Dutch: Het Driekanalenconcept: Het Effect op Voedingsinname Tijdens Ziekenhuisopname)
Brief Title: Three Channel Food Concept: the Effect Meal Service on Food Intake During Hospitalization
Status: Not yet recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 302653
Record Dates: First submitted 2024-03-05; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Nutrition Poor; Protein-Energy Malnutrition
MeSH Terms: conditions — Malnutrition; Protein-Energy Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- current in-hospital meal service: n=102 patients admitted to the Maastricht University Medical Centre+ (MUMC+) (surgical nursing wards) will be included.
  Interventions: Other: meal service
- old in-hospital meal service: This will be an historic control group (data already collected in the past)

INTERVENTIONS:
Other: meal service — We're not subjecting patients to an intervention, as we will evaluate the current in-hospital meal service. As the three channel food concept is standard of care, we're not subjecting patients to dietary or behavioral changes. We will compare the data to an historic control.
  Groups: current in-hospital meal service

SUMMARY:
The goal of this observational study is to assess food intake in hospitalized patients.

The present study will evaluate the impact of a novel in-hospital meal concept (three channel food concept) on total energy and protein intake, macronutrient distribution, and patient appreciation

Food intake will be assessed (as part of usual care) by weighing all leftovers (e.g. food that patients did not consume).

DETAILED DESCRIPTION:
There are various possible strategies to increase protein intake during hospitalization, such as providing more protein-rich foods, fortifying meals and/or food products, supplementation with oral nutritional supplements (ONS), and/or providing well-timed snacks. An appropriate in-hospital meal service is regarded as a key element of the strategy to minimize deterioration of the nutritional status. Conventional hospital meals, 3 main meals a day prepared by a central kitchen, are often low in protein and energy and are not appreciated by patients due to lack of taste, colour and flavour, resulting in inadequate food intake particularly protein intake. There are a number of avenues to improve nutritional intake, with type of meal service and existence of individual contact with catering staff, like mealtime assistance, as important factors. The MUMC+ has adapted it's in-hospital meal system and the present study will evaluate the impact of this novel in-hospital meal concept (three channel food concept) on total energy and protein intake, macronutrient distribution, and patient appreciation.

The aim of this study is to assess whether a novel in-hospital meal concept can effectively increase daily total protein and energy intake during hospitalization, when compared to a historic control.

ELIGIBILITY:
Inclusion Criteria:

* >18y
* Admitted to surgical nursing wards of MUMC+
* Expected hospital stay of at least 3 days

Exclusion Criteria:

* Receiving (par)enteral nutrition
* "NPO" (nil per os) policy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (>18y) admitted to surgery nursing wards of the Maastricht University Medical Centre+ (MUMC+).
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
total protein intake | during hospitalization (minimal 2days max 5days)
  total protein intake (g/kg/d)

SECONDARY OUTCOMES:
total energy intake | during hospitalization (minimal 2days max 5days)
  energy intake in kcal per day
macronutrient intake | during hospitalization (minimal 2days max 5days)
  carbohydrate, fat and protein intake (g/day)
Patient appreciation | during hospitalization (minimal 2days max 5days)
  Patient appreciation will be assessed using a question "what grade would you give the hospital food
Body weight upon hospital admission | upon hospital admission
  body weight in kilograms
Body height upon hospital admission | upon hospital admission
  body height in meters
reason hospital admission | upon hospital admission
  will be derived from electronical patient dossier

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Individual raw data can be shared upon reasonable request